CLINICAL TRIAL: NCT00657462
Title: Effect of Reminder Prompts on Utilization of the PAML Builder Application Features
Brief Title: Efficacy of the Pre-Admission Medication List (PAML) Builder Reminder Prompts
Acronym: PAMLTIPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Alexander Turchin, Senior Medical Informatician, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PAMLTIPS
Record Dates: First submitted 2008-04-09; First posted 2008-04-14 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Utilization of Software Application Features
Keywords: Medical Informatics Applications; Software; Utilization
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Receives the intervention (reminders displayed at the startup of the application) for both periods (period 1 and period 2) of the study.
  Interventions: Other: Reminders
- B (Active Comparator): Receives the intervention (reminders displayed at the application startup) only during the second period (period 2) of the study.
  Interventions: Other: Reminders

INTERVENTIONS:
Other: Reminders — Users of the PAML Builder application will receive reminders about three application features (copy/paste, audit trail, sort medications by class) at the startup of the application

SUMMARY:
This project will study whether reminder prompts increase PAML Builder application feature utilization.

DETAILED DESCRIPTION:
This project will study whether reminder prompts increase Pre-Admission Medication List (PAML) Builder application feature utilization. PAML Builder is an application designed and maintained by Partners Information Systems that assists clinicians in medication reconciliation - a process important for patient safety and quality of care. We have determined that several potentially helpful features of the application are not being utilized as frequently as had been expected. These features include:

1. copying the pre-admission medication list (PAML) to the clipboard
2. viewing the detailed audit trail of all changes made to the PAML
3. sorting the list of medications obtained from other electronic sources by therapeutic class.

Reminder prompts (sometimes referred to as "Tip of the Day") have been employed to increase user awareness of underutilized application features. However, anecdotally some users find them unhelpful and potentially irritating. It is therefore important to determine whether reminder prompts accomplish the stated task of increasing application feature utilization. This project will compare PAML Builder application feature utilization before and after a pilot rollout of reminder prompts to determine whether they should be implemented permanently.

ELIGIBILITY:
Inclusion Criteria:

* users of the PAML Builder application (physicians, nurses, pharmacists)

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 14122 (Actual)
Dates: Start 2008-04; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Difference in the change between combined frequency of utilization of all features promoted by the reminders per PAML built between the two arms from period 1 (intervention in one arm only) to period 2 (intervention in both arms). | The entire study period

SECONDARY OUTCOMES:
Difference in the change between frequencies of utilization of the individual features promoted by the reminders per PAML built between the two arms from period 1 (intervention in one arm only) to period 2 (intervention in both arms). | The entire study period
Difference in the change between combined frequency of utilization of all features promoted by the reminders per PAML built between the two arms from period 1 to period 2 by the users who were displayed the corresponding reminder. | The entire study period
Difference in the change between frequencies of utilization of the individual features promoted by the reminders per PAML built between the two arms from period 1 to period 2 by the users who were displayed the corresponding reminders. | The entire study period.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Turchin, MD, MS, Principal Investigator — Partners HealthCare; Carol Broverman, PhD, Principal Investigator — Partners HealthCare
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

REFERENCES:
- [Background] Poon EG, Blumenfeld B, Hamann C, Turchin A, Graydon-Baker E, McCarthy PC, Poikonen J, Mar P, Schnipper JL, Hallisey RK, Smith S, McCormack C, Paterno M, Coley CM, Karson A, Chueh HC, Van Putten C, Millar SG, Clapp M, Bhan I, Meyer GS, Gandhi TK, Broverman CA. Design and implementation of an application and associated services to support interdisciplinary medication reconciliation efforts at an integrated healthcare delivery network. J Am Med Inform Assoc. 2006 Nov-Dec;13(6):581-92. doi: 10.1197/jamia.M2142. PMID 17114640
- [Background] Turchin A, Gandhi TK, Coley CM, Shubina M, Broverman C. The use of electronic medication reconciliation to establish the predictors of validity of computerized medication records. Stud Health Technol Inform. 2007;129(Pt 2):1022-6. PMID 17911870